CLINICAL TRIAL: NCT03507907
Title: The Effects of Mulligan Mobilization Technique in Older Adults With Neck Pain: A Randomized Controlled, Double-Blind Study
Brief Title: The Effects of Mulligan Mobilization Technique in Older Adults With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018300
Record Dates: First submitted 2018-04-10; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Neck Pain
Keywords: neck pain; older adults; mobilization
MeSH Terms: conditions — Neck Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Mulligan mobilization techniques were applied to the older adults.
  Interventions: Other: Mulligan Mobilization for Study Group
- Control Group (Other): Conventional physiotherapy programs were applied to the older adults who included in control group.
  Interventions: Other: Conventional therapy for Control Group

INTERVENTIONS:
Other: Mulligan Mobilization for Study Group — Mulligan Mobilization techniques were applied to the older adults who included in study group.
  Arms: Study Group
Other: Conventional therapy for Control Group — Conventional therapy was applied to the older adults who included in control group.
  Arms: Control Group

SUMMARY:
When the literature is examined, there is study investigating the effect of mulligan mobilization technique on older adults with neck pain. This study aims to investigate the effect of mulligan mobilization technique on pain, range of motion, functional level, kinesiophobia, fear of movement, depression and quality of life in older adults with neck pain.

DETAILED DESCRIPTION:
Neck pain is common in older adults. There are a lot of approaches for treatment of neck pain such as soft tıssue mobilizations, electirical stimulations etc. Mulligan proposes mobilization with movement (MWM) technique for various musculoskeletal disorders. But there is no study related MWM for older adults with neck pain. The purpose of this study is to examine the effect of mulligan mobilization technique on pain, range of motion (ROM), functional level, kinesiophobia, depression and quality of life (QoL) in older adults with neck pain. The hypothesis of our study is MWM can be effective on ROM, kinesiophobia, depression and QoL in older adults with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing neck pain for at least 3 months,
* Having no neurological, rheumatological or musculoskeletal problems
* Having not taken any analgesic medication for neck pain for the last 3 months.

Exclusion Criteria:

* Neck pain originating from various pathologies
* Presence of cord compression,
* Vertebrobasilar artery insufficiency,
* Severe radiculopathy,
* Osteoporosis or osteopenia (t score>-1),
* Long-term use of anticoagulant or corticosteroid drugs,
* Patients who had received any treatment for their neck pain.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-10-14 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 5 months
  The severity of pain at rest and during activity was assessed by Visual Analogue Scale (VAS). Participants were questioned about their average pain over the last 4 weeks. They were asked to mark the severity of their pain on a 10-cm-long line where 0 represented no pain, and 10 stood for vicious pain

SECONDARY OUTCOMES:
Neck Disability Index | 5 months
  This scale was used to evaluate how the participants' daily life was influenced by their neck pain. Total score of the scale ranges from 0 to 35 and higher scores indicate higher levels of disability
Tampa Scale of Kinesiophobia | 5 months
  This scale was used to assess the patients' fear of pain or re-injury due to movement. It consists of 17 items and assesses various factors of fear/avoidance and injury/re-injury in several activities. Total score of the scale varies between 17 and 68 and higher scores represent higher levels of kinesiophobia.
Universal goniometer | 5 months
  A universal goniometer was used to assess the range of motion (ROM) of the cervical vertebrae. Cervical flexion, extension, right and left lateral flexion and right and left rotation movements were measured 3 times in active manner while the patients were in a comfortable sitting position. The average value of the measurements was recorded as ROM.
Beck Depression Inventory | 5 months
  Participants' level of depression was assessed using this scale that consists of 21 categories with 4 options in each. Each item has a score between 0 and 3 and total score varies from 0 to 63. Score ranges are interpreted as: 0-9 points = Minor depression, 10-16 points = Mild depression, 17-29 points = Moderate depression, and 30-63 points = Severe depression
Short Form-36 | 5 months
  This form was used to assess the quality of life (QoL) of the participants. This questionnaire is consisted of 36 questions that are categorized into 8 groups as following: physical role functioning, emotional role functioning, bodily pain, energy, social role functioning, mental health, and general health perception. Each category is scored on a 0-100 range, and higher scores indicate better QoL

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buyukturan O, Buyukturan B, Sas S, Kararti C, Ceylan I. The Effect of Mulligan Mobilization Technique in Older Adults with Neck Pain: A Randomized Controlled, Double-Blind Study. Pain Res Manag. 2018 May 15;2018:2856375. doi: 10.1155/2018/2856375. eCollection 2018. PMID 29861800